CLINICAL TRIAL: NCT00922311
Title: Aliskiren Combined With Losartan in Immunoglobulin A Nephropathy: an Open-label Pilot Study
Brief Title: Aliskiren for Proteinuric IgAN Despite Angiotensin Blockade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); United Christian Hospital (Other)
Responsible Party: Sydney CW Tang, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Novartis-ST-01
Record Dates: First submitted 2009-06-14; First posted 2009-06-17 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: IgA Nephropathy
Keywords: Proteinuria
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria | interventions — aliskiren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aliskiren (Experimental)
  Interventions: Drug: Aliskiren

INTERVENTIONS:
Drug: Aliskiren — Titrate from 150 mg daily to 300 mg daily
  Other Names: Rasilez

SUMMARY:
Study objective: To investigate the potential anti-proteinuric efficacy of aliskiren, a novel direct renin inhibitor (DRI), in addition to angiotensin receptor blocker (ARB) in immunoglobulin A nephropathy (IgAN) patients at risk of developing progressive renal failure.

DETAILED DESCRIPTION:
This will be an open-label pilot study in which IgAN patients with persistent proteinuria despite maximum dose of ARB treatment will be assigned to receive Aliskiren. There is the optional addition of other anti-hypertensive agents to achieve an optimal target blood pressure of <130/80 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 - 70 years of age
* Histologic diagnosis of IgA nephropathy
* Proteinuria > 1 g/day or UPC > 1 mg/mg or 113 mg/mmol at least twice
* Receiving treatment with the maximum dose of ARB for at least 3 months
* Patients who are willing to give written, informed consent

Exclusion Criteria:

* eGFR < 15 ml/min/1.73 sq.m
* UPC >5000 mg/g or 570 mg/mmol, or <500 mg/g or 57 mg/mmol
* Serum K+ > 5.2 mmol/L
* Presence of bilateral renal artery stenosis
* Presence of diabetes mellitus
* Renal histology showing pathologies other than IgAN
* Known allergy to ARB or DRI
* Patients on ARB/ACEi combination within 12 weeks of randomization
* Concurrent treatment with corticosteroids, Nsaid, or immunosuppressant
* Patients with connective tissue disease or obstructive uropathy
* Patients with malignancy or conditions severely limiting life expectancy
* Female who are pregnant or intending to conceive
* Female of child-bearing age unwilling to practice contraception
* Patients who are unable to give informed consent
* Patients simultaneously participating in another study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change of urine protein excretion rate | 6 months

SECONDARY OUTCOMES:
Changes in serum creatinine, eGFR, serum potassium and albumin | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sydney CW Tang, MD, Principal Investigator — The University of Hong Kong
Locations (2):
- China (2):
  - Department of Medicine, The University of Hong Kong, Hong Kong
  - Queen Mary Hospital, Hong Kong

REFERENCES:
- [Derived] Tang SC, Lin M, Tam S, Au WS, Ma MK, Yap DY, Ho YW, Lai KN. Aliskiren combined with losartan in immunoglobulin A nephropathy: an open-labeled pilot study. Nephrol Dial Transplant. 2012 Feb;27(2):613-8. doi: 10.1093/ndt/gfr349. Epub 2011 Jun 16. PMID 21680850